CLINICAL TRIAL: NCT07384364
Title: A Prospective, Single-Arm, Observational Case Series Evaluation of the Impact of Robotic Spinal Mobilization on Functional Mobility, Axial Rigidity, Chronic Back Pain, and Sleep Quality in Community-Dwelling Adults With Parkinson's Disease
Brief Title: Observational Study Evaluating Robotic Spinal Mobilization in 16 Parkinson's Disease Participants. The Study Recorded Changes in Mobility, Sit-to-stand Performance, and Pain Scores After a 2-week Intervention With the BackHug Device.
Status: Completed | Type: Observational
Sponsor: Pacla Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-PD-2025-01
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson Disease; Axial Rigidity; Robotic Spinal Mobilization; Functional Mobility; Pain; Sleep quality
MeSH Terms: conditions — Parkinson Disease; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this completed observational pilot study was to evaluate the immediate and short-term clinical effects of robotic spinal mobilization on motor and non-motor symptoms in community-dwelling adults with Parkinson's Disease (PD). Specifically, the study aimed to determine if the mechanical release of axial rigidity correlates with measurable improvements in functional mobility, postural stability, and symptom burden.

A cohort of 16 participants (Hoehn and Yahr Stages 1-3) attended four 40-minute therapy sessions using the BackHug device over a two-week period. The device utilizes 26 robotic fingers to deliver targeted deep-tissue mobilization to the paraspinal muscles and intervertebral joints.

Researchers assessed outcomes using a repeated-measures design. Functional mobility and strength were measured immediately before and after sessions to capture acute therapeutic effects. Subjective metrics for chronic back pain and sleep quality were monitored longitudinally to assess cumulative benefits. The study provides preliminary data on the feasibility and efficacy of non-invasive mechanical mobilization as an adjunct therapy for PD.

DETAILED DESCRIPTION:
Study Rationale and Background: Axial rigidity is a cardinal motor feature of Parkinson's Disease (PD) that contributes significantly to gait impairment, balance dysfunction, and chronic pain. Unlike appendicular symptoms, axial symptoms often show limited response to standard dopaminergic medication. This study investigated the utility of the BackHug robotic device to mechanically mobilize the thoracic and lumbar spine, evaluating the hypothesis that reducing axial stiffness improves systemic mobility.

Technical Description of the Intervention: The BackHug device is an automated spinal mobilization system featuring 26 independent robotic therapeutic heads. The mechanism employs real-time load sensing to adapt pressure to the user's spinal curvature. Participants received a standardized 40-minute protocol targeting the neck, shoulders, thoracic, and lumbar spine. Treatment intensity was personalized to user tolerance via the device's control app.

Quality Assurance and Data Validation Plan: To ensure data integrity and minimize bias in this observational setting, the following quality assurance procedures were implemented:

* Administrator Qualifications: All functional assessments were administered by HCPC-registered physiotherapists trained in standard PD assessment protocols (e.g., TUG, STS) to ensure inter-rater reliability.
* Source Data Verification: Primary functional data was recorded on standardized paper Assessment Forms (source documents) at the point of care. These were subsequently verified against the electronic study database.
* Video Verification: Where participant consent was granted, video recordings of functional tests were utilized as source data to cross-verify the accuracy of timed metrics (e.g., confirming gait speed to the nearest millisecond).
* Data Consistency Checks: The data management system employed logic checks during entry to flag out-of-range values (e.g., age outside 18-75, VAS scores outside 0-10) for immediate review against clinician notes.

Data Management and Missing Data

Data Dictionary: All variables were defined according to standard clinical scales (e.g., Visual Analog Scale 0-10 cm; Likert Scale 1-5).

Handling of Missing Data: The study adhered to a Per-Protocol analysis. Missing data points resulting from missed sessions or incomplete assessments were documented in the study log but excluded from the final efficacy calculation for that specific endpoint. No data imputation methods were used.

Statistical Analysis Plan

Sample Size Assessment: As a pilot observational case series, the sample size (N=16) was determined based on feasibility and the capacity of the single-center clinical facility. The objective was to generate effect size estimates and standard deviation data sufficient to power a future randomized controlled trial (RCT).

Descriptive Statistics: Baseline demographics (Age, Gender, Disease Duration) were summarized using means and standard deviations.

Efficacy Analysis: The primary analytical method compared Pre-Intervention vs. Post-Intervention scores to determine the percentage change in performance. Paired t-tests were employed to assess the statistical significance of acute and longitudinal changes in functional mobility and strength.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Confirmed clinical diagnosis of Parkinson's Disease.
* Disease Severity: Hoehn and Yahr Scale Stage 3 or below (indicating mild to moderate disability with preserved postural reflexes).
* Functional Mobility: Ability to walk independently for approximately 5 minutes. Use of walking poles is permitted; reliance on a walking frame (Zimmer frame) or wheelchair excludes participation.
* Consent: Willing and able to provide informed consent and attend all four scheduled therapy sessions.

Exclusion Criteria:

* Spinal & Bone Pathology: Diagnosis of spinal malignancy (benign or malignant tumors), active spinal infection (e.g., tuberculosis), severe congenital defects (dysplasia), metabolic bone disease (e.g., severe osteomalacia), or currently healing spinal fractures/dislocations.
* Inflammatory Conditions: Severe Rheumatoid Arthritis or other inflammatory arthritides causing potential spinal instability.
* Neurological Contraindications (Non-PD): Evidence of spinal cord compression, spinal cord damage, or Cauda Equina syndrome.
* Vascular & Hematological Risks: History of aortic dysfunction (e.g., abdominal aortic aneurysm, blood clot), severe haemophilia, or unmanaged bleeding disorders.
* Other: Current pregnancy; History of active cancer (excluding localized squamous cell carcinoma); Recent spinal surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort was selected from a community-dwelling population in Edinburgh, United Kingdom. Recruitment was conducted at a single specialist physiotherapy centre (The Manual Therapy Clinic) through patient database referrals and local outreach. The population comprised individuals with a confirmed diagnosis of Parkinson's Disease who were living independently in the community and actively seeking non-pharmacological management for motor symptoms
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Functional Mobility (3-Meter Timed Up and Go Test) | Baseline (Session 1) and Post-Intervention (Session 4, approximately 2 weeks later).
  Functional mobility is assessed using the 3-Meter Timed Up and Go (TUG) test. Participants are timed (in seconds) as they rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. This test evaluates gait speed, balance, and functional agility. A decrease in time indicates an improvement in mobility.

SECONDARY OUTCOMES:
Change in Subjective Back Pain Intensity (Visual Analog Scale) | Baseline (Session 1) and Post-Intervention (Session 4, approximately 2 weeks later).
  Participants self-report their current level of back pain intensity using a Visual Analog Scale (VAS) ranging from 0 to 10.
  0 = No Pain 10 = Worst Possible Pain A decrease in the score indicates a reduction in pain intensity.
Change in Self-Reported Sleep Quality | Baseline (Session 1) and Post-Intervention (Session 4, approximately 2 weeks later).
  Participants rate their overall sleep quality using a numerical rating scale from 0 to 5.
  0 = Very Poor Sleep 5 = Excellent Sleep An increase in the score indicates an improvement in sleep quality and restoration.

CONTACTS AND LOCATIONS:
Locations (1):
- The Manual Therapy Clinic, Edinburgh, Scotland, United Kingdom